CLINICAL TRIAL: NCT02047045
Title: Effect Comparison of Electro-acupuncture and Prucalopride for Severe Chronic Constipation: a Multi-center Noninferiority Randomized Controlled Trial
Brief Title: Effect Comparison of Electro-acupuncture and Prucalopride for Severe Chronic Constipation: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Zhishun, Dean of Acupuncture Department of Guang'anmen Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012BAI24B01SCC
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-02

CONDITIONS: Constipation
Keywords: severe chronic constipation; randomized controlled; electro-acupuncture; prucalopride
MeSH Terms: conditions — Constipation | interventions — Acupuncture Therapy; prucalopride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electro-acupuncture (Experimental): Electro-acupuncture at bilateral ST25, SP14 ,and ST37. Patients will be treated once per day for 30 min, 5 times/week for the first 2 weeks, and 3 times/week for the next 6 weeks.
  Interventions: Procedure: acupuncture
- Prucalopride (Active Comparator): Prucalopride Succinate taken orally, 2mg/day in the morning before breakfast
  Interventions: Drug: Prucalopride

INTERVENTIONS:
Procedure: acupuncture — Electro-acupuncture at bilateral ST25, SP14 ,and ST37. Patients will be treated once per day for 30 minutes, 5 times/week for the first 2 weeks and 3 times/week for the next 6 weeks. Each treatment cycle will include 28 sessions for continuous 8 weeks.
  Other Names: eletro-acupuncture
  Arms: Electro-acupuncture
Drug: Prucalopride — Prucalopride Succinate will be taken orally at the dose of 2mg/day in the morning before breakfast. Each treatment cycle will be given for continuous 32 weeks.
  Other Names: serotonin 5-HT(4) receptor agonist
  Arms: Prucalopride

SUMMARY:
This trial is primarily aimed to compare the effect and safety of electro-acupuncture and prucalopride for severe chronic constipation: if the short-term effect of electro-acupuncture is no inferior to prucalopride? Besides, the investigators will also mainly confirm the superiority of electro-acupuncture: if the effect of electro-acupuncture can last for 3~6 months? Then, assess the patients' acceptance of electro-acupuncture.

DETAILED DESCRIPTION:
Study design: this trial is a multi-central randomized controlled trial which contains 14 centers. Random sequences will be generated by the clinical evaluating center of China Academy of Chinese Medical Sciences. Subjects are patients who have severe chronic constipation.

Sample size evaluation: Sample size will be based on the proportion of patients having mean complete spontaneous bowel movements (CSBMs) no less than 3 times per week. The proportion is 31.67% in our phase I clinical trial by using electro-acupuncture, and 30.9% in another trial by using prucalopride.The total sample size is 560.

Periods and primary outcome: participants will be assessed at baseline for 2 weeks, treated for 8 weeks, and followed up for 24 weeks. Primary outcome is the proportion of patients having mean CSBMs/week no less than 3 times over the latter 6-week treatment.

Quality control: the study is a randomized controlled trial; participants were included strictly; evaluators and statisticians are blinded; quality control officers of 3 different levels will supervise this trial.

Data management: this trial will use the Remote Dara Capture (RDC) system for data entering and Data Verification Plan (DVP) for data examining.

Statistical analysis: Intention-To-Treat (ITT) analysis will be used in this study. One-sided test (non-inferiority) will be used for testing the primary outcomes; meanwhile, two-sided test will be used for evaluating other outcomes. A P value equal to or less than 0.05 is considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. meeting Rome Ⅲ criteria for diagnosing functional constipation;
2. severe chronic constipation (two or fewer CSBMs per week for more than 3 months）;
3. the weekly mean CSBMs are no more than 2 times during the 2-week baseline
4. aged from 18 to 75 years old
5. no use of drugs for constipation (emergency treatments should be excepted) during at least 2 weeks before enrollment; no acupuncture treatment for constipation in the previous 1 month; never joined any other trial in progress;
6. volunteered to join this research and signed the informed consent

Exclusion Criteria:

1. irritable bowel syndrome, organic constipation or secondary constipation caused by endocrine, metabolic, nervous, postoperative diseases, or by drugs;
2. mushy stool or watery stool are showed more than once during baseline when defecating spontaneously without any laxative (Bristol stool type 6 or 7);
3. history of pelvic floor dysfunction;
4. taking medicine in progress which can induce constipation;
5. severe hemorrhoid or anal fissure;
6. constipation with serious cardiovascular, hepatic or renal diseases, cognitive dysfunction, abdominal aortic aneurysm or hepatosplenomegaly, aphasia, mental disorders, or illness which affects the cooperation for examination and treatment;
7. women in gestation or lactation period;
8. blood coagulation disorders or using anticoagulants regularly such as Warfarin and Heparin;
9. cardiac pacemaker carrier.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Ph.D, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: Yes
Data sharing study protocol, informed consent form, and statistical analysis plan are in the supplementary digital files with the clinical report. For statistical code and data sets, proposals should be directed to yanshiyan0927@sina.com, and requestors need to sign a data access agreement, if approved.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within six months after the publication of the clinical report
Access Criteria: For statistical code and data sets, proposals should be directed to yanshiyan0927@sina.com, and requestors need to sign a data access agreement, if approved.

REFERENCES:
- [Background] Liu B, Wang Y, Wu J, Mo Q, Wang W, He L, Yan S, Liu Z. Effect of electroacupuncture versus prucalopride for severe chronic constipation: protocol of a multi-centre, non-inferiority, randomised controlled trial. BMC Complement Altern Med. 2014 Jul 23;14:260. doi: 10.1186/1472-6882-14-260. PMID 25055821
- [Result] Liu B, Wu J, Yan S, Zhou K, He L, Fang J, Fu W, Li N, Su T, Sun J, Zhang W, Yue Z, Zhang H, Zhao J, Zhou Z, Song H, Wang J, Liu L, Wang L, Lv X, Yang X, Liu Y, Sun Y, Wang Y, Qin Z, Zhou J, Liu Z. Electroacupuncture vs Prucalopride for Severe Chronic Constipation: A Multicenter, Randomized, Controlled, Noninferiority Trial. Am J Gastroenterol. 2021 May 1;116(5):1024-1035. doi: 10.14309/ajg.0000000000001050. PMID 33273258
- [Derived] Gao S, Zhu L, Yao H, Fang J, Liu Z. Effect of electroacupuncture versus prucalopride for ultra-severe chronic constipation: Secondary analysis of a randomized controlled trial. Integr Med Res. 2026 Mar;15(1):101253. doi: 10.1016/j.imr.2025.101253. Epub 2025 Sep 12. PMID 41080507

RESULTS

PARTICIPANT FLOW:
Groups:
- Prucalopride: Prucalopride Succinate taken orally, 2mg/day in the morning before breakfast
  Prucalopride: Prucalopride Succinate will be taken orally at the dose of 2mg/day in the morning before breakfast. Each treatment cycle will be given for continuous 8 weeks.
Period: Baseline
Arm/Group | Electro-acupuncture | Prucalopride
Started | 280 | 280
Completed | 277 | 278
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2
Period: Treatment Period (8 Weeks )
Arm/Group | Electro-acupuncture | Prucalopride
Started | 277 | 278
Completed | 266 | 263
Not Completed | 11 | 15
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 3 | 5
Not completed — moved far away out of work | 3 | 0
Not completed — no reason was given | 1 | 0
Not completed — refused to take drugs | 0 | 5
Not completed — for safety considerations | 0 | 1
Period: Follow-up Period (24 Weeks)
Arm/Group | Electro-acupuncture | Prucalopride
Started | 266 | 263
Completed | 265 | 262
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population was the recruited patients with baseline data. We recruited 560 participants (280 for each group) in total; however, 3 participants from EA group and 2 from prucalopride group withdrew their informed consents with no baseline data. Therefore, they were not included in the baseline analysis.
Groups:
- Electro-acupuncture: Electro-acupuncture (EA) at bilateral ST25, SP14 ,and ST37. Additionally, bilateral BL33 was used for severe straining if any; DU20 and DU24 were used for patients with anxiety and depression if any.
  EA treatment was lasted for 30 min, and EA treatment was taken 5 times/week for the first 2 weeks, and 3 times/week for the next 6 weeks. Each treatment cycle will include 28 sessions for continuous 8 weeks.
  After the EA treatment is stopped, the participants will be followed up for 24 weeks.
- Prucalopride: Prucalopride Succinate was taken orally, 2mg/day in the morning before breakfast for continuous 8 weeks.
  Participants took electrocardiograph (ECG) at day 7 of the 8th week. Participants would take prucalopride for additional 24 weeks if no significant ECG changes (such as prolonged QT intervals) showed.
- Total: Total of all reporting groups
Arm/Group | Electro-acupuncture | Prucalopride | Total
Number analyzed (Participants) | 277 | 278 | 555
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.06 (16.12) | 45.79 (16.00) | 45.93 (16.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 224 | 446
  Male | 55 | 54 | 109
Race/Ethnicity, Customized [Number; unit: participants]
  Han | 270 | 275 | 545
  Others | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  China | 277 | 278 | 555

OUTCOME MEASURES:

1. Primary Outcome: the Proportion of Participants With ≥3 Mean Weekly CSBMs Over Weeks 3-8
Description: Abbreviation: CSBMs, complete spontaneous bowel movements. Calculation method: First, the mean weekly CSBMs of each patient were calculated over weeks 3-8. Second, we got the number of patients with 3 or more mean weekly CSMBs. Third, we got the proportion of participants through dividing that number by the total cases at baseline, and multiplying by 100%.
  Assessing time frame: the latter 6 weeks of treatment (weeks 3-8).
Time Frame: over weeks 3-8 (the latter 6-week treatment)
Population: We recruited 560 participants (280 for each group) in total; however, 3 participants from EA group and 2 from prucalopride group withdrew their informed consents. Therefore, they were not included in the baseline analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
percentage of participants | 36.2 | 37.8

2. Secondary Outcome: the Proportion of Participants With ≥3 Mean Weekly CSBMs Over Weeks 1-2, 11-12, 15-16, 19-20, 31-32.
Description: Abbreviation: CSBMs, complete spontaneous bowel movements. Calculation method: First, the mean weekly CSBMs of each patient were calculated over weeks 1-2, 11-12, 15-16, 19-20, 31-32. Second, we got the number of patients with 3 or more mean weekly CSMBs. Third, we got the proportion of participants through dividing that number by the total cases at baseline, and multiplying by 100%.
  Assessing time frame: weeks 1-2, 11-12, 15-16, 19-20, 31-32.
Time Frame: over weeks 1-2, 11-12, 15-16, 19-20, 31-32.
Population: We recruited 560 participants (280 for each group) in total; however, 3 participants from EA group and 2 from prucalopride group withdrew their informed consents. Therefore, they were not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
percentage of participants
  weeks 1-2 | 27.1 | 33.8
  weeks 11-12 | 38.3 | 43.2
  weeks 15-16 | 38.0 | 41.0
  weeks 19-20 | 35.7 | 42.1
  weeks 31-32 | 37.6 | 38.5

3. Secondary Outcome: the Proportion of Participants With ≥1 Increase in Mean Weekly CSBMs From Baseline Over Weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Description: Abbreviation: CSBMs, complete spontaneous bowel movements. Calculation method: First, the increase in mean weekly CSBMs of each patient from baseline were calculated over weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32. Second, we got the number of patients with ≥1 increase in the mean weekly CSMBs from baseline. Third, we got the proportion of participants through dividing that number by the total cases at baseline, and multiplying by 100%.
  Assessing time frame: weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Time Frame: over weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
percentage of participants
  weeks 1-2 | 49.5 | 61.5
  weeks 3-8 | 66.4 | 63.3
  weeks 11-12 | 63.5 | 63.7
  weeks 15-16 | 65.7 | 66.2
  weeks 19-20 | 61.4 | 64.0
  weeks 31-32 | 61.0 | 61.5

4. Secondary Outcome: Mean Weekly CSBMs and Its Change From Baseline Over Weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Time Frame: over weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: bowel movements
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
bowel movements
  weeks 1-2 | 1.27 [1.17 to 1.38] | 1.78 [1.66 to 1.89]
  weeks 3-8 | 1.96 [1.86 to 2.06] | 1.97 [1.87 to 2.08]
  weeks 11-12 | 2.00 [1.90 to 2.10] | 2.01 [1.90 to 2.12]
  weeks 15-16 | 1.93 [1.82 to 2.03] | 2.07 [1.95 to 2.18]
  weeks 19-20 | 1.90 [1.80 to 2.00] | 2.00 [1.89 to 2.11]
  weeks 31-32 | 1.94 [1.83 to 2.05] | 1.99 [1.89 to 2.10]

5. Secondary Outcome: Mean Weekly SBMs and Its Change From Baseline Over Weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Time Frame: over weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: bowel movements
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
bowel movements
  weeks 1-2 | 1.85 [1.72 to 1.98] | 2.91 [2.78 to 3.03]
  weeks 3-8 | 2.13 [2.03 to 2.24] | 2.60 [2.49 to 2.70]
  weeks 11-12 | 1.87 [1.76 to 1.97] | 2.43 [2.33 to 2.54]
  weeks 15-16 | 1.65 [1.53 to 1.76] | 2.38 [2.28 to 2.49]
  weeks 19-20 | 1.59 [1.48 to 1.70] | 2.33 [2.22 to 2.44]
  weeks 31-32 | 1.50 [1.38 to 1.62] | 2.24 [2.13 to 2.36]

6. Secondary Outcome: the Change From Baseline in Mean Score of Stool Consistency for Each SBM Over Weeks 1-2 and 3-8.
Description: The change from baseline in the mean score of stool consistency of each SBM over weeks 1-2 and weeks 3-8. Assessing time: baseline, weeks 1-2 and weeks 3-8. Patients will self-report their stool consistency of each SBM according to the 7-type Bristol Stool Form Scale (scored by 1 to 7 respectively). Type 1: Separate hard lumps, like nuts (hard to pass); Type 2: Sausage-shaped, but lumpy; Type 3: Like a sausage but with cracks on its surface; Type 4: Like a sausage or snake, smooth and soft; Type 5: Soft blobs with clear cut edges (passed easily); Type 6: Fluffy pieces with ragged edges, a mushy stool; Type 7: Watery, no solid pieces. Entirely liquid.
  Type 3 and 4 were deemed as a normal stool.
Time Frame: over weeks 1-2, 3-8.
Population: The number of participants providing data of stool consistency was 270 in EA group and 266 in prucalopride group.
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 270 | 266
score
  weeks 1-2 | 0.48 [-0.08 to 1.13] | 0.67 [0.06 to 1.38]
  weeks 3-8 | 0.78 [0.12 to 1.40] | 0.74 [0.17 to 1.42]

7. Secondary Outcome: the Change From Baseline in Mean Score of Straining for Each SBM Over Weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Description: The change from baseline in the mean score of straining of each SBM over weeks 1-2, 3-8, 9-12, 9-16, 9-20, 9-32. Assessing time: baseline, weeks 1-2, 3-8, 9-12, 9-16, 9-20, 9-32. Patients will self-report their straining degree of each SBM in the defecation diaries according to the following scale. 0 = not difficult; 1 = a little difficult, need some straining to defecate; 2 = difficult, need straining to defecate; 3 = very difficult, need hard straining to defecate. Higher scores mean a worse outcome.
Time Frame: over weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Population: The number of participants providing data of straining was 271 in EA group and 266 in prucalopride group over weeks 1-2/3-8; The number of participants providing data of straining was 264 in EA group and 261 in prucalopride group over weeks 11-12/15-16/19-20/31-32.
Measure: Median (Inter-Quartile Range); unit: score
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 271 | 266
score
  weeks 1-2 | -0.33 [-0.83 to 0.00] | -0.52 [-1.00 to 0.00]
  week 3-8 | -0.54 [-0.98 to -0.15] | -0.63 [-1.00 to -0.13]
  weeks 11-12: number analyzed (Participants) | 264 | 261
  weeks 11-12 | -0.60 [-1.13 to -0.14] | -0.58 [-1.14 to 0.00]
  weeks 15-16: number analyzed (Participants) | 264 | 261
  weeks 15-16 | -0.59 [-1.16 to -0.13] | -0.57 [-1.13 to 0.00]
  weeks 19-20: number analyzed (Participants) | 264 | 261
  weeks 19-20 | -0.67 [-1.20 to -0.17] | -0.67 [-1.18 to 0.00]
  weeks 31-32: number analyzed (Participants) | 264 | 261
  weeks 31-32 | -0.67 [-1.29 to -0.13] | -0.67 [-1.24 to 0.00]

8. Secondary Outcome: Time to the First CSBMs
Description: Abbreviation: CSBMs, complete spontaneous bowel movements. Time to the first CSBMs was counted by days. Rescue medicine or other measurements for constipation is not allowed to be used 48 hours before and after the first treatment for evaluating the time to the first complete spontaneous bowel movement. Participants were assessed after the first treatment until they having their first CSBMs.
Time Frame: from the time of their first treatment to the time they having their first CSBMs
Population: The number of participants providing data of time to the first CSBMs was 272 in EA group and 266 in prucalopride group.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 272 | 266
days | 4 [0 to 7] | 5 [0 to 7]

9. Secondary Outcome: Change From Baseline in Mean Score of Patient Assessment of Constipation Quality of Life
Description: The change from baseline of the score of Patient Assessment of Constipation Quality of Life (PAC-QOL) at week 4 and week 8. PAC-QOL is a self-report questionnaire to evaluate the quality of life in patients with constipation, which was distributed by Mapi Research Trust in France. This questionnaire contains 28 items including 4 basic parts of physical discomfort, worries and concerns, psychosocial discomfort, and satisfaction. We use the Chinese version in our trial. Assessing point: baseline, week 4 and week 8. The score of PAC-QOL ranged from 1 to 5 (1 indicates no discomfort or feeling very satisfied, 5 indicates extreme severity and always appears or feeling very dissatisfied).
Time Frame: week 4 and week 8
Population: The number of participants providing data of PAC-QOL was 261 in EA group and 260 in prucalopride group at week 4; The number of participants providing data of PAC-QOL was 261 in EA group and 257 in prucalopride group at week 8.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 261 | 260
score
  week 4 | -0.71 (0.64) | -0.72 (0.69)
  week 8: number analyzed (Participants) | 261 | 257
  week 8 | -1.09 (0.79) | -1.00 (0.78)

10. Other Pre Specified Outcome: Proportion of Patients Using Rescue Medicine Over Weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Time Frame: over weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Measure: Number; unit: percentage of participants
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
percentage of participants
  weeks 1-2 | 13.72 | 7.91
  weeks 3-8 | 19.49 | 17.99
  weeks 11-12 | 9.75 | 6.83
  weeks 15-16 | 10.47 | 7.19
  weeks 19-20 | 10.83 | 5.76
  weeks 31-32 | 10.11 | 6.47

11. Other Pre Specified Outcome: Average Dosage of Bisacodyl Used Weekly Over Weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Time Frame: over weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Measure: Median (Inter-Quartile Range); unit: tablet
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
tablet
  weeks 1-2 | 0.75 [0.50 to 1.00] | 0.50 [0.50 to 2.50]
  weeks 3-8 | 0.17 [0.17 to 0.33] | 0.67 [0.33 to 1.50]
  weeks 11-12 | 0.50 [0.50 to 1.00] | 0.75 [0.50 to 2.00]
  weeks 15-16 | 0.50 [0.50 to 1.00] | 0.50 [0.50 to 1.50]
  weeks 19-20 | 0.50 [0.50 to 1.00] | 1.00 [0.50 to 1.25]
  weeks 31-32 | 0.50 [0.50 to 1.00] | 1.00 [0.50 to 2.00]

12. Other Pre Specified Outcome: Average Dosage of Glycerine Enema Used Weekly Over Weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Time Frame: over weeks 1-2, 3-8, 11-12, 15-16, 19-20, 31-32.
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
ml
  weeks 1-2 | 40.00 [20.00 to 55.00] | 55.00 [40.00 to 60.00]
  weeks 3-8 | 18.33 [11.67 to 30.00] | 18.33 [10.00 to 35.00]
  weeks 11-12 | 30.00 [20.00 to 67.50] | 20.00 [10.00 to 52.50]
  weeks 15-16 | 55.00 [30.00 to 80.00] | 22.50 [20.00 to 50.00]
  weeks 19-20 | 52.50 [30.00 to 80.00] | 45.00 [25.00 to 52.50]
  weeks 31-32 | 55.00 [30.00 to 55.00] | 37.50 [20.00 to 55.00]

13. Post Hoc Outcome: the Proportion of Overall CSBM Responders Over Weeks 1-8
Description: A weekly CSBM responder was defined as a patient who had ≥3 CSBMs for a given week and an increase from baseline of ≥1 CSBM for that same week. An overall CSBM responder was a patient who was a weekly CSBM responder for at least 6 of the 8 treatment weeks (75%).
Time Frame: over weeks 1-8
Measure: Number; unit: percentage of participants
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
percentage of participants | 24.91 | 25.54

14. Post Hoc Outcome: the Proportion of Sustained CSBM Responder Over Weeks 1-8
Time Frame: over weeks 1-8
Measure: Number; unit: percentage of participants
Arm/Group | Electro-acupuncture | Prucalopride
Number analyzed (Participants) | 277 | 278
percentage of participants | 24.91 | 24.46

ADVERSE EVENTS:
Time Frame: the whole study period (34 weeks, from week -2 to week 32)
Description: We recruited 560 participants (280 for each group) in total; however, 3 participants from EA group and 2 from prucalopride group withdrew their informed consents. Therefore, they were not included in the analysis.
Arm/Group | Electro-acupuncture | Prucalopride
Serious Adverse Events (participants affected / at risk) | 1/277 | 0/278
Other Adverse Events (participants affected / at risk) | 49/277 | 123/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Electro-acupuncture (N=277) | Prucalopride (N=278)
Cardiac surgery due to myocardial infarction (Cardiac disorders) | 1 | 0 — This severe adverse event is unrelated to EA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Electro-acupuncture (N=277) | Prucalopride (N=278)
Nausea (Gastrointestinal disorders) | 1 | 22
Abdominal Pain (Gastrointestinal disorders) | 4 | 38
Fever (General disorders) | 2 | 4
Faint (General disorders) | 1 | 5
Diarrhea (Gastrointestinal disorders) | 4 | 36
Bloating (Gastrointestinal disorders) | 1 | 3
Cold (General disorders) | 10 | 25
Headache (General disorders) | 4 | 34
Dizziness (General disorders) | 2 | 20
Palpitation (Cardiac disorders) | 0 | 12
Blood-stained stools due to diarrhea (Gastrointestinal disorders) | 0 | 1
High uric acid (Renal and urinary disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Aches (Musculoskeletal and connective tissue disorders) | 0 | 1
Sense of hunger (Gastrointestinal disorders) | 0 | 1
Scapulohumeral periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot sprain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck and shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spondylosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Local hematoma (Skin and subcutaneous tissue disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Fear or nervous (Psychiatric disorders) | 1 | 0
Dry mouth (Nervous system disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 0 | 1
Sprain (Musculoskeletal and connective tissue disorders) | 1 | 1
Emesis (Gastrointestinal disorders) | 0 | 2
Hyperplasia of mammary glands (Reproductive system and breast disorders) | 1 | 0
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper limb numbness (Nervous system disorders) | 1 | 0
Pyelonephritis (Renal and urinary disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Empyrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Arthrolithisis (Immune system disorders) | 1 | 0
Dysmenorrhea (Reproductive system and breast disorders) | 1 | 2
Distention in head (General disorders) | 0 | 1
Leg Hurt (Musculoskeletal and connective tissue disorders) | 0 | 1
Stomachache (Gastrointestinal disorders) | 1 | 4
Knee Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Knee joint pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Chest distress and short of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Elevated blood pressure (General disorders) | 1 | 0
Toothache (General disorders) | 1 | 1
Pharyngalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Soreness of waist (Musculoskeletal and connective tissue disorders) | 0 | 1
Low back pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Lumbar disc herniation (Musculoskeletal and connective tissue disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Wrist sprain (Musculoskeletal and connective tissue disorders) | 0 | 1
Premature menstruation (Reproductive system and breast disorders) | 2 | 0
Fatty liver (Hepatobiliary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes